CLINICAL TRIAL: NCT06358911
Title: A Clinical Study for the Effect of 4th Generation Poly Amido Amine Dendrimer (PAMAM-COOH) Desensitizing Agent on Post-Bleaching Hypersensitivity and Shade Stability of Patients Subjected to Bleaching Treatment.
Brief Title: A Clinical Study for the Effect of 4th Generation Poly AmidoAmine Dendrimer on Post-Bleaching Hypersensitivity and Shade Stability
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: FDASU-RecID022001
Record Dates: First submitted 2024-04-06; First posted 2024-04-11 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Tooth Hypersensitivity
Keywords: Dental Bleaching; Shade Stability
MeSH Terms: conditions — Dentin Sensitivity | interventions — Durapatite

STUDY DESIGN:
Intervention Model Description: This clinical study will be conducted to evaluate the effect of using 4th generation Poly amido amine dendrimer (PAMAM-COOH) as a desensitizing agent and compared with three different commercially available desensitizing materials: 3% potassium nitrate and 0.11% fluoride (Ultra EZ), as described by manufacturer, Casein-phosphopeptide-amorphous calcium phosphate with F, (MI paste plusTm), and Hydroxyapatite, Fluoride and Xylitol, Hydroxyapatite and F (ReminPro), on:
  1. Long-term Post-bleaching hypersensitivity.
  2. Long-term Post-bleaching shade stability. For Patients treated with 40% hydrogen-peroxide bleaching agent.
Who Masked: Participant, Outcomes Assessor
Masking Description: This clinical trail was a double blinded trail in which the participant and outcome assessor were blinded to allocation, thus the participant was unaware of which experimental material had been assigned to him/her. Also outcome assessors were blinded to the treatment that each participant had received
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Poly amido amine dendrimer (PAMAM)'s desensitizing agent (Experimental): Fourth generation with COOH terminal functional group, colorless liquid. PAMAM-succinamic acid dendrimer, 1,4-diaminobutane core, generation 4 solution. 10 wt.% in water.
  The application of PAMAM 30 min according to previous studies
  Interventions: Other: Poly amido amine dendrimer (PAMAM)
- Manufacturer's desensitizing agent, Ultra EZ (Experimental): 3% potassium nitrate and 0.11% fluoride (Ultra EZ), gel The application of manufacturer recommended desensitizing agent for 1hrs
  Interventions: Other: Manufacturer's desensitizing agent, Ultra EZ
- MI paste plus, desensitizing agent (Experimental): Casein-phosphopeptide-amorphous calcium phosphate with Fluoride, topical tooth cream.
  Gel contains pure water,D-sorbitol,glycerol,Carboxymethylcellulose Sodium, casein phosphopeptide amorphous calcium phosphate,propylene glycol, titanium dioxide, Silicon dioxide, Sodium Saccharin,Phosphoric acid, butyl P-hydroxy-benzoate, and ethyl hydroxyl benzoate
  The application of MI paste plus according to manufacturer instructions, 3minutes
  Interventions: Other: MI paste plus, desensitizing agent
- Hydroxyapatite and F (ReminPro), desensitizing agent (Experimental): Hydroxyapatite, Fluoride and Xylitol, water-based cream The application of Hydroxyapatite and F (ReminPro) according to manufacturer instructions, 3minutes
  Interventions: Other: Hydroxyapatite and F (ReminPro), desensitizing agent

INTERVENTIONS:
Other: Poly amido amine dendrimer (PAMAM) — Desensitizing agents was applied once after the bleaching procedure,as follows:
  1-Bleaching/PAMAM group, patients received bleaching followed by the application of PAMAM for 30 minutes according to previous studies.
  Arms: Poly amido amine dendrimer (PAMAM)'s desensitizing agent
Other: Manufacturer's desensitizing agent, Ultra EZ — Desensitizing agents was applied once after the bleaching procedure, as follows:
  2-Control group, where patients received hydrogen peroxide in-office bleaching followed by the application of manufacturer recommended desensitizing agent ( Ultra EZ) once for 60 minutes.
  Arms: Manufacturer's desensitizing agent, Ultra EZ
Other: MI paste plus, desensitizing agent — Desensitizing agents was applied once after the bleaching procedure, as follows:
  3-Bleaching/MI Paste Plus group, patients received bleaching followed by the application of MI paste plus according to the manufacturer's instructions once for 3 minutes.
  Arms: MI paste plus, desensitizing agent
Other: Hydroxyapatite and F (ReminPro), desensitizing agent — Desensitizing agents was applied once after the bleaching procedure, as follows:
  4-Bleaching/Hydroxyapatite and F (ReminPro), patients received bleaching followed by the application of Hydroxyapatite and F (ReminPro) according to the manufacturer's instructions once for 3 minutes
  Arms: Hydroxyapatite and F (ReminPro), desensitizing agent

SUMMARY:
This study assessed the impact of four desensitizing agents on both color stability and dental sensitivity following a bleaching procedure, spanning from the 24-hour to the 1-year follow-up assessment periods.

DETAILED DESCRIPTION:
Dental bleaching is a temporary treatment with potential adverse effects on dental sensitivity post-procedure. Therefore, the study aimed to evaluate dental color stability and sensitivity over a one-year period following bleaching, utilizing one of four desensitizing agents: PAMAM, MI Paste Plus, Hydroxyapatite and F (ReminPro), and Ultra EZ. The selection of the desensitizing agent was based on a predetermined randomization sequence generated in Microsoft Excel. Color stability was objectively assessed through spectrophotometric analysis, while subjective evaluation was conducted using the Vita Classic shade guide by two external observers not involved in the procedure. Dental sensitivity levels were tracked at various intervals using a visual analogue scale. Baseline measurements for both sensitivity and color stability were taken before the bleaching procedure, with subsequent evaluations at 24 hours, 3 days, 1 week, 1 month, 3 months, 6 months, 9 months, and 1 year post-bleaching. The study involved 60 patients from Ain Shams University seeking dental whitening treatment, divided into four groups based on the randomization sequence.

ELIGIBILITY:
Inclusion Criteria:

Male and female patients will be selected according to the following inclusion criteria:

* Participants should have their entire upper and lower teeth, from right first premolar to left first premolar, present and sound, without restorations or periodontal disease.
* Teeth have never been bleached before.
* The participants are required to have low-caries index.
* Teeth should have a Vita-color shade of A2 or darker.
* Cooperative behavior patient and medically free.
* Patient ages between 18 to 40 years old.

Exclusion Criteria:

* Serious medically compromised patients.
* Smoking, alcoholism.
* Hypersensitivity to the agents used in the study.
* Lactated, pregnant patients.
* Patients have serious oral diseases, as acute necrotizing gingivitis, acute gingiva stomatitis, or undergoing orthodontic treatment.
* Patients with dental enamel cracks.
* Patients who had previous bleaching treatments

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-11-13 (Actual); Primary Completion 2023-08-05 (Actual); Study Completion 2023-09-10 (Actual)

PRIMARY OUTCOMES:
Post-bleaching dental hypersensitivity | 24 hours 3 days, 7 days, 1 month, 3 months, 6 months, 9 months and one year post treatment
  Assessment will be carried out by a visual analogue scale (VAS), from 0 (no tooth sensitivity at all) to 10 (intolerable pain). Air blast stimulus will be used and will be applied on the tooth at distance of 0.5-1 cm for 2 seconds by the maximum power of the compressed air jet from the dental unit. Then sensitivity was measured before bleaching (baseline) and at each follow up period, 24 hours, 3 days, 7 days, 3 months, 6 months, 9 months, and one year post treatment
Shade stability | 24 hours 3 days, 7 days, 1 month, 3 months, 6 months, 9 months and one year post treatment
  Assesment was carried out using Vita Easy shade V . Two measurements were taken for each tooth from the upper right canine to the upper left canine, and same for the lower arch. For light condition standardization, all shade measurements were carried out under natural daylight the clinic lights with the dental unit light away from the patient. The shade of each tooth was recorded as well as the values of L, a, and b. The shade of the upper two centrals was confirmed using Vita Classical shade guide.
  Shade assesment was carried out before bleaching and at each follow up periods, 24 hours, 3 days, 7 days, 3 months, 6 months, 9 months, and one year post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Farid MS Al Askary, Professor, Study Director — Ain Shams University
Locations (1):
- Faculty of Dentistry - Ain Shams University, Cairo, El Weili, Egypt

IPD SHARING:
Plan to Share IPD: No